CLINICAL TRIAL: NCT06786481
Title: Effect of Foot Massage Performed to the Mother After Post-Bırth on Breastfeedıng Success, Sleep Qualıty and Neonatal Stress: a Randomızed Controlled Study
Brief Title: Effect of Foot Massage Performed to the Mother After Bırth on Breastfeedıng Success, Sleep Qualıty and Newborn Stress
Status: Active, not recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Melek Nur KEÇELİ (Other)
Responsible Party: Sponsor-Investigator, Melek Nur KEÇELİ, Principal Investigator, Kahramanmaras Sutcu Imam University
Organization: Kahramanmaras Sutcu Imam University (Other)
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Supportive Care
Other Study IDs: KahramanmaraşSIUA
Record Dates: First submitted 2024-09-26; First posted 2025-01-22 (Actual); Last update posted 2025-01-22 (Actual); Status verified 2025-01

CONDITIONS: Postpartum Women
Keywords: reflexology massage, breastfeeding success, sleep quality, newborn stress
MeSH Terms: conditions — Sleep Initiation and Maintenance Disorders | interventions — Milnacipran; Massage; Lactation

STUDY DESIGN:
Intervention Model Description: Parallel asigment
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (1):
- Experimental (Experimental): Before starting the foot massage, the client is informed about the number, duration and time of the session. The average interview time with the patients in the experimental group will be 15-20 minutes. The first interview with the women in the experimental group will be held at any time after the birth when the woman feels well. Before the application, the researcher washes and dries her hands and warms them appropriately by massaging with baby oil and facilitates the process. First, a three-minute general massage is performed to prepare the feet, and then the correct points for each foot are massaged for 10 minutes. 'Introductory Information Form', "LATCH Breastfeeding Diagnostic Measurement Tool", "Newborn Stress Scale" and "Pittsburgh Sleep Quality Index (PSQI)" forms will be filled. The woman's address and telephone details will be taken to meet again.
  Interventions: Behavioral: Educational with milnacipran; Behavioral: Locally Directed Therapy

INTERVENTIONS:
Behavioral: Educational with milnacipran — Before starting the foot massage, the client is informed about the number, duration and time of the session. The average interview time with the patients in the experimental group will be 15-20 minutes. The first interview with the women in the experimental group will be held at any time after the birth when the woman feels well. Before the application, the researcher washes and dries her hands and warms them appropriately by massaging with baby oil and facilitates the process. First, a three-minute general massage is performed to prepare the feet, and then the correct points for each foot are massaged for 10 minutes. 'Introductory Information Form', "LATCH Breastfeeding Diagnostic Measurement Tool", "Newborn Stress Scale" and "Pittsburgh Sleep Quality Index (PSQI)" forms will be filled. The woman's address and telephone details will be taken to meet again.
Behavioral: Locally Directed Therapy — Before starting the foot massage, the client is informed about the number, duration and time of the session. The average interview time with the patients in the experimental group will be 15-20 minutes. The first interview with the women in the experimental group will be held at any time after the birth when the woman feels well. Before the application, the researcher washes and dries her hands and warms them appropriately by massaging with baby oil and facilitates the process. First, a three-minute general massage is performed to prepare the feet, and then the correct points for each foot are massaged for 10 minutes. 'Introductory Information Form', "LATCH Breastfeeding Diagnostic Measurement Tool", "Newborn Stress Scale" and "Pittsburgh Sleep Quality Index (PSQI)" forms will be filled. The woman's address and telephone details will be taken to meet again.
  Other Names: kortizol; massage; breastfeeding

SUMMARY:
Aim: To Reveal The Effect Of Foot Massage Performed To The Mother After Bırth On Breastfeedıng Success, Sleep Qualıty And Newborn Stress Material and Method: This randomized controlled trial was conducted with 70 people (35 experimental, 35 control) in a public hospital in Kahramanmaraş.

DETAILED DESCRIPTION:
: Aim: To Reveal The Effect Of Foot Massage Performed To The Mother After Bırth On Breastfeedıng Success, Sleep Qualıty And Newborn Stress Material and Method: This randomized controlled trial was conducted with 70 people (35 experimental, 35 control) in a public hospital in Kahramanmaraş.

In the first stage, the researcher participants were informed about the purpose of the researcher and the questionnaire, and their consent was obtained for participation in the study.

In the second stage, Before starting the foot massage, the client will be informed about the number of sessions, their duration, and when they will be held. The average interview time for the patients in the experimental group will be 15-20 minutes. The first interview with the women in the experimental group will be held at any time after birth when the woman feels well. Before the application, the researcher washes and dries her hands, and massages them with baby oil to warm them up properly and facilitate the process. First, a three-minute general massage is given to prepare the feet, and then the correct points are massaged for 10 minutes for each foot. The "Introductory Information Form", "LATCH Breastfeeding Diagnostic Measurement Tool", "Neonatal Stress Scale", and "Pittsburgh Sleep Quality Index (PSQI)" forms related to the study will be filled out. The woman's address and telephone information will be obtained in order to meet again.

ELIGIBILITY:
Inclusion Criteria:

* Literate,

  * Communicative,
  * Poor sleep status (with a global score of ≧5 on the PSQI,
  * Patients who volunteer to participate in the study,
  * Minimum and maximum gestational age of 37 and 42 weeks,
  * No psychological disorder,
  * Low-risk singleton pregnancy,
  * Good foot health (cuts, burns, fungus, warts, etc.)
  * No sensitivity to touch or massage.

Exclusion Criteria:

* Those who wish to withdraw from the study, • Patients with deficiencies or errors in any of the forms used to collect data will be removed from the study.

Sex: Female | Healthy Volunteers: Yes
Age Groups: Child, Adult, Older Adult
Enrollment: 70 (Estimated)
Dates: Start 2025-01-01 (Actual); Primary Completion 2025-07-30 (Estimated); Study Completion 2025-08-30 (Estimated)

PRIMARY OUTCOMES:
LATCH | 30 day
  It was developed by Jensen and Wallace in 1994 in order to perform breastfeeding assessment objectively and systematically, to identify breastfeeding problems, to establish a common language among healthcare professionals and to be used in studies. It is similar to the apgar score system in terms of scoring method. This measurement tool consists of five assessment items. The word LATCH is a combination of the first letters of the English equivalents of these items.
Neonatal Stress Scale | 30 day
  The neonatal stress scale developed by Ceylan and Bolışık consists of a total of 24 items in 3-point Likert type. The scale items include 8 subgroups including facial expression, body colour, respiration, activity level, comfort, muscle tone, extremities and posture and each subgroup is evaluated between 0-2 points in scoring. A minimum score of 0 and a maximum score of 16 points are obtained from the scale. As the score increases, the stress level of the baby increases simultaneously.

CONTACTS AND LOCATIONS:
Locations (1):
- Melek Nur Keçeli, Kahramanmaraş, Turkey (Türkiye)

IPD SHARING:
Plan to Share IPD: No